CLINICAL TRIAL: NCT04811339
Title: Pilot and Randomized, Controlled Studies to Assess Stool Frequency of COVID + Patients Treated With Oral Bismuth Subsalicylate (Pepto-Bismol): SABER-C and Lite-SABER-C (Specific Administration of Bismuth for Early Recovery of COVID-19)
Brief Title: Studies of COVID-19 Patients Treated With Oral Bismuth Subsalicylate (Pepto-Bismol)
Acronym: SABER-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Bruce Yacyshyn, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SABER-C 20.0636
Record Dates: First submitted 2021-03-20; First posted 2021-03-23 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Diarrhea; COVID-19
MeSH Terms: conditions — Diarrhea; COVID-19 | interventions — Tablets; Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Intervention Model Description: Open label trial of Bismuth subsalicylate (10 patients) followed by a second, placebo controlled study (50 patients) for mild to moderate COVID-19+ patients.
Who Masked: Outcomes Assessor
Masking Description: Member of research team not involved in patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Open label BSS (Experimental): All patients will be assigned to the treatment group for the first 10 patients treated with open label BSS.
  Interventions: Drug: Bismuth Subsalicylate 262 milligram (mg) Oral Tablet, Chewable
- Randomized BSS or Placebo (Placebo Comparator): The Subsequent 50 patients will be randomized to either placebo or BSS. The patients will be assigned by envelope containing a symbol for either active drug or placebo (or other suitable randomization event) by a member of the research team not directly involved in the clinical trial.
  Interventions: Drug: Bismuth Subsalicylate 262 milligram (mg) Oral Tablet, Chewable; Other: Placebo oral tablet without BSS

INTERVENTIONS:
Drug: Bismuth Subsalicylate 262 milligram (mg) Oral Tablet, Chewable — Pepto bismol (bismuth subsalicylate)
  Other Names: Pepto Bismol
Other: Placebo oral tablet without BSS — Placebo Tablet made by P & G to contain everything except active ingredient ( BSS)
  Arms: Randomized BSS or Placebo

SUMMARY:
The Center for Disease Control (CDC) and World Health Organization (WHO) have deemed the COVID-19 virus a global pandemic of unprecedented severity in modern times. In 2019, this novel Coronavirus (COVID-19) emerged from the Asian continent and has now caused upwards of 1million deaths and over 6 million infections globally. Currently, the estimated global economic impact is over 5 Trillion dollars. Understanding the host response to pathogens, specifically the cellular and humoral responses, has played an important role in new non-antibiotic therapies. Bismuth subsalicylate (Pepto-Bismol) has a potential role in the clearance and/or recurrence of enteric viral infections.

DETAILED DESCRIPTION:
Readily available over-the-counter (OTC) medication for symptomatic relief and appropriate oral hydration can be health saving measures of great convenience for those affected by enteric bacterial and viral infections. BSS is a non-proprietary monograph product that is available in the USA and abroad, over-the-counter (OTC). Of all OTC medications for traveller's diarrhea (TD), bismuth subsalicylate (BSS) has the greatest antimicrobial activity against pathogenic bacteria .BSS has also exhibited significant inhibition on viral invasion of host cells and viral efficacy. Both BSS and bismuth oxychloride (BiOCl, which is formed in the stomach after ingestion of BSS) at low concentration (0.004-0.13mg/mL) significantly reduced norovirus (NoV) RNA levels, suggesting an in vivo antiviral mechanism. BSS has also been shown to have antiviral activity since it inhibited replication of 4 strains of rotavirus in tissue culture cells and caused a dose-dependent reduction in the growth of several enteric viruses.

Historically, BSS has been indicated and effectively used for the treatment of TD or enteric infection, mainly when vomiting occurs. Although the safety and efficacy of BSS is well known, some of the research done with BSS resides within the industry and have not been published. We have recently completed an extensive meta-analysis using unpublished clinical studies regarding BSS safety and efficacy. Meta-analyses of randomized controlled clinical trials were performed with studies specifically designed to capture prevention of manifestation and relief of diarrhea.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, patients must meet the following criteria: Ability to provide written or remote informed consent (telephone and DocuSign) Ability to comply with study requirements, Men or women 18 to 85 years of age, inclusive Current diagnosis of an initial occurrence of non-severe, non-complicated COV+ infection as defined by:

* Presence COVID-19 in the saliva using point of care (POC) Qualitative real time - polymerase chain reaction (QRT- PCR) assay.
* Management in an outpatient (i.e., non-hospital) or inpatient setting NOT on a ventilator.
* Alert and awake
* Able to chew the study drug completely.
* Women should fulfill one of the following criteria:
* Answer in the affirmative that "they are not or could not be pregnant"
* Post-menopausal; either amenorrhea ≥12 months or follicle stimulating hormone >20 mIU/mL (milli-International units)
* Surgically sterile; hysterectomy, bilateral oophorectomy, or tubal ligation.
* Women of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception from Screening through the 21 Day visit, per Section 10.2.

Standard of care COVID-19 treatment is acceptable.

Exclusion Criteria:

Patients with any of the following will be excluded from admission into the study:

* Existence of an intra-abdominal abscess, enteric fistula, or symptomatic bowel obstruction
* History of allergy to salicylates.
* History of short gut syndrome, active ulcer or recent history of GI bleeding or melena.
* Systemic chemotherapy for the treatment of cancer during the 60 days prior to consent or planned during the study
* Active use of remdesivir.
* vaccination for COVID within 30 days.
* Current use of drugs that control diarrhea or affect peristalsis (e.g., loperamide. Opiates can be used in hospitalized patients and with outpatients if they are prescribed to a patient), or any anticipated use during the study
* Active drug, chemical, or alcohol dependency as determined by Investigator through history or urine toxicology screen
* Enrollment in any other investigational drug or device study known to interfere with Pepto bismol (bismuth subsalicylate) within the GI tract, within 30 days prior to Randomization (Day 1) or within 5 half-lives of the last dose of the previous investigational compound, whichever is longer. Vaccines are not exclusionary as they do not interfere with the mechanism of the study drug.
* Severe acute illness unrelated to COVID-19
* Pregnant, breast-feeding, or considering becoming pregnant during the study
* Planned hospitalization or surgery during the study
* Any medical, psychiatric, social, or other circumstances that may interfere with study compliance, completion, or accurate assessment of study outcomes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Yacyshyn, MD, Principal Investigator — Adjunct Professor Systems Physiology and Pharmacology University of Cincinnati
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yacyshyn MB, Collins J, Chua M, Siegwald A, Yacyshyn S, Briones-Pryor V, Yacyshyn B. Feasibility study of Bismuth Subsalicylate (BSS) as an addition to standard of care for COVID-19 therapy. Curr Ther Res Clin Exp. 2022;96:100667. doi: 10.1016/j.curtheres.2022.100667. Epub 2022 Mar 30. No abstract available. PMID 35370296
- [Background] Brum JM, Gibb RD, Ramsey DL, Balan G, Yacyshyn BR. Systematic Review and Meta-Analyses Assessment of the Clinical Efficacy of Bismuth Subsalicylate for Prevention and Treatment of Infectious Diarrhea. Dig Dis Sci. 2021 Jul;66(7):2323-2335. doi: 10.1007/s10620-020-06509-7. Epub 2020 Aug 8. PMID 32772204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The open label feasibility arm started Oct 2020 and completed Feb 2021 at University of Louisville Hospitals. First patient consented and received drug was on Oct 27 2020, last patient Feb 20 2021. This was pre vaccine environment. Public availability of vaccine in Kentucky was March of 2021. 19 patients received drug with only 10 patients completing therapy. Placebo controlled study (50 patients) was cancelled. If started a new study will be entered in Clinical.Trials.gov
Pre-assignment Details: 19 patients received drug. 9 patients received some Bismuth Subsalicylate (BSS), 10 patients completed 3 days of BSS therapy. All was done in pre-vaccine environment. 25 patients consented received no drug.
Groups:
- BSS Open Label: 10 patients will be treated with open label BSS and complete the 3 day therapy.
  Open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
  10 patients need to complete this feasibility arm
- Consented Only No Drug: 25 consented but received no drug. Most were early on in the recruitment of patients.
- SOC Control Group - Cancelled: This part of the study has been cancelled. The Subsequent 50 patients would have been randomized to either placebo or BSS. However, the placebo was confiscated at the border and became outdated and we could not use.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
Period: Overall Study
Arm/Group | BSS Open Label | Consented Only No Drug | SOC Control Group - Cancelled
Started (19 patients received some BSS. 10 completed and 9 did not complete) | 19 (19 patients were given BSS.) | 25 (No drug given) | 0
Complete 3 Days of BSS (To complete BSS therapy, patients also needed to provide 3 days of saliva for SARS-CoV2 testing, record three days of bowel movements and record and score (between 0-3) 5 symptoms : cough, headache, fatigue, shortness of breath and anosmia ( loss of smell)) | 10 | 0 | 0
Completed | 10 (10 persons did complete all requirements of taking BSS and providing all samples and answering all questions) | 0 | 0
Not Completed | 9 | 25 | 0
Not completed — lack of transportation not wanting to return | 4 | 8 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Inconclusive saliva SARS CoV2 test (3X) | 1 | 0 | 0
Not completed — Negative primary or secondary salivary SARS-CoV2 test | 0 | 6 | 0
Not completed — Medications. Standard of Care medications were changing rapidly Protocol needed constant amending | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Transferred to ICU for non-COVID-19 related problem | 0 | 1 | 0
Not completed — Early on Nurse/Physician communication issue | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: 44 persons needed to be consented in order to reach 10 persons who would complete therapy and all sample collections. In the pre vaccine environment and earlier in the pandemic problems with retention and ever changing standard of care environments and just patient and staff generalized fear made it more difficult than anticipated to reach just 10 persons who would complete BSS oral therapy.
Groups:
- Open Label BSS Therapy -Completed: All patients will be assigned to the treatment group for the first 10 patients treated with open label BSS.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
  10 who completed 3 day therapy and provided all samples
- Open Label BSS Therapy - Those Who DID NOT Complete: 9 patients who got some BSS - but did not complete 3 day therapy
- Open Label - BSS Therapy No BSS Given: Those 25 patients who consented but received no BSS therapy.
- Cancelled Placebo-control & BSS Arm: The Subsequent 50 patients would have been randomized to either placebo or BSS. The patients will be assigned by envelope containing a symbol for either active drug or placebo (or other suitable randomization event) by a member of the research team not directly involved in the clinical trial.
  We could not recruit due to confiscation and expiration of placebo.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
- Total: Total of all reporting groups
Arm/Group | Open Label BSS Therapy -Completed | Open Label BSS Therapy - Those Who DID NOT Complete | Open Label - BSS Therapy No BSS Given | Cancelled Placebo-control & BSS Arm | Total
Number analyzed (Participants) | 10 | 9 | 25 | 0 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 6 | 5 | 15 |  | 26
  >=65 years | 4 | 4 | 10 |  | 18
Age, Continuous [Mean (Standard Deviation); unit: year] | 52.70 (21.79) | 65.22 (8.84) | 60.6 (14.58) |  | 59.75 (15.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 11 |  | 19
  Male | 5 | 6 | 14 |  | 25
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was taken from Electronic Health Records (EHR)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 |  | 0
    Asian | 0 | 0 | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 |  | 1
    Black or African American | 2 | 2 | 7 |  | 11
    White | 8 | 7 | 17 |  | 32
    More than one race | 0 | 0 | 0 |  | 0
    Unknown or Not Reported | 0 | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 25 |  | 44
Number of pre-existing Comorbidities [Mean (Full Range); unit: Comorbidities] — Only patients that were consented and received any BSS had this parameter collected. Population: Only those patients who received any BSS had this parameter collected. Those that were consented but received no drug - only had basic demographic information collected
  Comorbidities
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 3.7 [0 to 10] | 4.7 [3 to 8] |  |  | 4.2 [0 to 10]
Number of pre-existing home medications [Mean (Full Range); unit: Home medications] — Population: Only those who received any BSS had this measure collected. Those consented but who received not drug did not have this parameter collected
  Home medications
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 3.8 [0 to 13] | 4.8 [1 to 10] |  |  | 4.4 [0 to 13]
Number of COVID-19 symptom days prior to study entry [Mean (Full Range); unit: days] — Days were used counted prior to date of consent. Asymptomatic -patients had data represented as 0. Population: Only those who received any BSS had this parameter collected. Those consented but had received no BSS did not have this parameter collected
  days
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 8.5 [0 to 19] | 9.1 [0 to 30] |  |  | 10.6 [5 to 30]
Number of COVID-19 morbidities [Mean (Full Range); unit: COVID-19 related morbidities] — Population: Only those patients who received drug had this parameter measured. Those who were consented but received no drug did not have this parameter measured
  COVID-19 related morbidities
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 3.5 [0 to 9] | 2.4 [1 to 4] |  |  | 3 [0 to 9]
Baseline/Day1 5 symptom score [Mean (Full Range); unit: Scores on a Scale] — The 5 symptom composite score was generated using 5 symptoms: Cough, Headache, Fatigue, Shortness of Breath, and Anosmia (no smell). Each symptom was scored from 0 - 3. Zero was not affected, 1 was little affected, 2 moderately affected, 3 severely affected. A composite score was generated using the sum from each symptoms score. The minimum composite score was 0 and the maximum was 15. Higher composite score equalled greater patient perceived Covid symptomatic impact on how they were feeling. A lower composite score represented that a patient felt they had fewer and less severe symptoms. Population: Only patients who received any BSS had this parameter measured. Those consented but who did not receive BSS did not have this parameter recorded
  Scores on a Scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 3.8 [1 to 9] | 3.2 [0 to 11] |  |  | 3.5 [0 to 11]
Baseline/Day1 3 symptom score [Mean (Full Range); unit: Scores on scale] — The 3 symptom composite score was generated from 3 symptoms: Cough, Headache and Fatigue Each symptom was scored as such: 0 was not affected, 1 was little affected, 2 moderately affected, 3 severely affected. A composite score was generated using the score given for each individual symptom. The minimum composite score could be 0 and maximum most symptomatic composite score would be 9. A higher composite score represented that a patient felt more and greater symptomatic effects from Covid Infection. The lower the score, the patient would report fewer and less severe symptoms due to Covid. Population: Parameter recorded only for those patients who received any BSS. Those patients consented who did not receive BSS did not have this parameter recorded
  Scores on scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 2.4 [0 to 5] | 2.1 [0 to 8] |  |  | 2.4 [0 to 8]
Baseline Health Score [Mean (Full Range); unit: scores on scale] — The Baseline Health score (BHS) was a composite generated from 3 different parameters.
  (1) Number of COVID-19 symptoms; actual patient range recorded was 0-5. (2) Number of preexisting comorbidities; actual patient range recorded was 0 - 10. (3) Number of COVID-19 related morbidities; actual patient range recorded was 0 - 9. Theoretical BHS composite score range is 0 - 24. A higher score at baseline represented greater impact of Covid infection on the patient prior to medication. A lower score represented a less severe Covid impact on the patient prior to medication. Population: This score was calculated for those patients who received any drug. Those patients who consented but did not receive any medication did not have this score calculated.
  scores on scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 19
    (all) | 9.3 [5 to 18] | 9.1 [4 to 14] |  |  | 9.2 [4 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Measure of Daily Stool Frequency for Patients With COVID Treated With Bismuth
Description: Number of bowel movements recorded over the 3 day study. Baseline (BL) /day1 + Day 2 + Day 3
Time Frame: 3 days
Population: Data from 10 completed patients.
Measure: Mean (Standard Error); unit: bowel movements
Groups:
- Open Label BSS Completed Patients: All patients will be assigned to the treatment group for the first 10 patients treated with open label BSS.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
- SOC Control Group: The Subsequent 50 patients will be randomized to either placebo or BSS. The patients will be assigned by envelope containing a symbol for either active drug or placebo (or other suitable randomization event) by a member of the research team not directly involved in the clinical trial.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
Arm/Group | Open Label BSS Completed Patients | SOC Control Group
Number analyzed (Participants) | 10 | 0
bowel movements | 3 (0.5) |

2. Secondary Outcome: Salivary SARS-CoV2 Day 3 Status Using Reverse-transcription Loop-mediated Isothermal Amplification (RT-LAMP)
Description: Salivary SARS-CoV2 measured daily. The final outcome is SARS-CoV2 status on day 3. Clearance of SARS-CoV2 ( a negative salivary SARS-CoV2 RT-LAMP test). or Remained SARS-CoV2+ ( a positive salivary SARS-CoV2. RT-LAMP test)
Time Frame: Day 3 - or 48 hours after starting BSS
Population: These 10 patients completed BSS therapy and provided 3 days of saliva for RT-LAMP testing for presence or absence of SARS-CoV2
Measure: Count of Participants; unit: Participants
Groups:
- Open Label BSS Therapy -Completed: Patients who completed BSS therapy
- Cancelled SOC Control Group: This next arm of study cancelled due to placebo being impounded and then expired. The Subsequent 50 patients were to be randomized to either placebo or BSS arms. The patients will be assigned by envelope containing a symbol for either active drug or placebo (or other suitable randomization event) by a member of the research team not directly involved in the clinical trial.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
Arm/Group | Open Label BSS Therapy -Completed | Cancelled SOC Control Group
Number analyzed (Participants) | 10 | 0
Participants
  Those who cleared salivary SARS-CoV2 | 5 | 0
  Those who remained salivary SARS-CoV2 positive | 5 | 0

3. Post Hoc Outcome: Day 3 Composite 5 Symptom Score
Description: The 5 symptom composite score was generated from 5 symptoms: Cough, Headache, Fatigue, Shortness of Breath, and Anosmia (no smell). Each symptom was scored as such: 0 was not affected, 1 was little affected, 2 moderately affected, 3 severely affected. A composite score was generated using the score given for each individual symptom, ie. the sum of symptomatic score of Cough + symptomatic score of Headache + symptomatic score of Fatigue + symptomatic score of Shortness of Breath + symptomatic score of anosmia. The maximum and most symptomatic composite score could be 15 each day. The minimum score could be 0. This score was calculated calculated for BL/day1, day 2 and day 3 . This outcome is the composite 5 symptom score on day 3.
Time Frame: The score was taken at BL (baseline)/day 1, Day 2 ( 24 hours after BSS started ) and Day 3 (48 hours after BSS started). This Outcome is Day 3 score.
Population: Those 10 patients who completed BSS open label therapy
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Open Label BSS Therapy -Completed | Cancelled SOC Control Group
Number analyzed (Participants) | 10 | 0
score on a scale | 2.9 [0 to 7] |

4. Post Hoc Outcome: Day 3 Composite 3 Symptom Score
Description: The 3 symptom composite score was generated from 3 symptoms: Cough, Headache, and Fatigue. Each symptom was scored as such: 0 was not affected, 1 was little affected, 2 moderately affected, 3 severely affected. A composite score was generated using the score given for each individual symptom, ie. the sum of symptomatic score of Cough + symptomatic score of Headache + symptomatic score of Fatigue. The maximum and most symptomatic composite score could be 9 each day. The minimum score could be 0 . This score was calculated calculated for BL/day1, day 2 and day 3 . This outcome is the composite 3 symptom score on day 3.
Time Frame: This is the day 3 composite score
Population: These 10 patients completed the open label BSS study
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Open Label BSS Therapy -Completed | Cancelled SOC Control Group
Number analyzed (Participants) | 10 | 0
score on a scale | 1.4 [0 to 4] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 3 days of the BSS study.
Description: Patients were asked to report any side effects
Groups:
- Cancelled SOC Control Group: This group was cancelled. The Subsequent 50 patients would have been randomized to either placebo or BSS. The patients will be assigned by envelope containing a symbol for either active drug or placebo (or other suitable randomization event) by a member of the research team not directly involved in the clinical trial.
  open label BSS (pepto Bismol): Pepto bismol (bismuth subsalicylate)
Arm/Group | Open Label BSS Therapy -Completed | Open Label BSS Therapy - Those Who DID NOT Complete | Cancelled SOC Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 3/9 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label BSS Therapy -Completed (N=10) | Open Label BSS Therapy - Those Who DID NOT Complete (N=9) | Cancelled SOC Control Group (N=0)
Abdominal bloating (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 — The patients felt bloated or let the coordinators know they had abdominal discomfort

LIMITATIONS AND CAVEATS:
1. Changing Standard of Care.
2. Patients, floor nurses and coordinators did not always keep track of number of pills taken.
3. For better compliance, we needed to decrease number of pills/day from 24 or 8 per day.
4. Transportation after discharge and sample collection needed to be optimized.
5. There was surprising difficulty in recruiting and maintaining patients in the trial during the first year, prior to general vaccine availability. 25 patients consented and never received drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT04811339/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04811339/ICF_001.pdf